CLINICAL TRIAL: NCT02342613
Title: Adoptive Immunotherapy Utilizing Activated Marrow Infiltrating Lymphocytes Derived From Patients With Bone Marrow Relapse of Hematologic Malignancies After Allogeneic Hematopoietic Cell Transplantation Using Post-Transplantation Cyclophosphamide Graft-Versus-Host Disease Prophylaxis.
Brief Title: Adoptive Immunotherapy With Activated Marrow Infiltrating Lymphocytes and Cyclophosphamide Graft-Versus-Host Disease Prophylaxis in Patients With Relapse of Hematologic Malignancies After Allogeneic Hematopoietic Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1484; IRB00039074 (Other: JHM IRB); P01CA153962 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hematologic Malignancies; Graft-Versus-Host Disease
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MILs treatment (Experimental): Patients treated with the activated PTCy-MILs
  Interventions: Biological: Activated PTCy-MILs

INTERVENTIONS:
Biological: Activated PTCy-MILs — The activated PTCy-MILs will be infused through standard blood tubing containing a 170-260 micron filter without an additional leukoreduction filter into a central IV site. Each of the bags will be infused at a rate of approximately 10 ml per minute. The IV line will be flushed with normal saline immediately after completion of PTCy-MILs infusion to ensure that all product has been infused into the patient.

SUMMARY:
This Phase 1 clinical study is designed to examine the safety and feasibility of using anti-CD3/CD28 activated marrow infiltrating lymphocytes (MILs) as treatment of relapse after allogeneic hematopoietic cell transplantation (alloHCT) for patients with hematologic malignancies with bone marrow involvement of their relapsed disease. These MILs will be derived from the bone marrow of the relapsed patient who had previously received post-transplantation cyclophosphamide (PTCy) as graft-versus-host disease (GVHD) prophylaxis (PTCy-MILs). A bone marrow aspiration will be performed on the patient to collect ~200ml of marrow for ex vivo expansion. During this expansion process, T cells will be activated and expanded by co-stimulation with anti-CD3/anti-CD28 monoclonal antibodies covalently attached to super-paramagnetic microbeads. Patients will be treated with salvage therapy while this ex vivo expansion is ongoing. After the simultaneous salvage therapy and ex vivo expansion, the activated PTCy-MILs will be reinfused. Patients will be monitored with the primary objective being the feasibility of expanding to targeted dose levels activated PTCy-MILs that do not cause grade III-IV acute GVHD within the first 90 days after PTCy-MIL infusion.

DETAILED DESCRIPTION:
Primary Objectives:

1. Feasibility of generating activated PTCy-MILs in patients with relapsed disease involving the bone marrow.
2. Toxicity of PTCy-MILs, specifically the rate of grade III-IV acute GVHD within the first 90 days after PTCy-MIL infusion.

Secondary Objectives

1. Determination of an optimal safe dose for PTCy-MILs.
2. Immunologic characterization of the PTCy-MIL product before and after expansion.
3. Immune reconstitution after treatment with PTCy-MILs.
4. Incidence and severity of chronic GVHD.
5. Clinical responses (complete remissions, partial remissions, stable disease) as measured by criteria specific for the particular disease type.
6. Progression-free and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Bone marrow relapse of a hematologic malignancy ≥6 months after alloHCT using PTCy
* Donor CD3+ chimerism ≥ 30% measured in peripheral blood or bone marrow
* ECOG performance status ≤ 2 or Karnofsky performance scale ≥ 70%.
* Off all immunosuppressive drugs for 2 weeks prior to the PTCy-MILs collection.
* Expectation of ability to safely undergo salvage treatment appropriate for the patient's malignant disease type as determined by the treating hematologist/ oncologist.

Exclusion Criteria:

* Most recent alloHCT not utilizing PTCy.
* Active GVHD requiring treatment.
* Immunosuppression use within 28 days of PTCy-MIL infusion if prior grade II-IV acute GVHD.
* Creatinine ≥ 2.5, total bilirubin > 3 times the upper limit of normal (ULN), or AST/ALT > 3 times the ULN.
* HIV-1/2 or HTLV-1/2 positivity.
* Life expectancy ≤ 90 days even with aggressive treatment, as determined by the treating hematologist/oncologist, which would preclude assessment of toxicity of PTCy-MILs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of generating activated marrow infiltrating lymphocytes (MILs) from participants previously treated with post-transplantation cyclophosphamide (PTCy) (PTCy-MILs) who have relapsed disease involving the bone marrow | 90 days
  Feasibility is measured as the number of participants who achieve: 1) The successful obtaining of PTCy-MILs; 2) The expansion of PTCy-MILs to at least 70% of the assigned dose level; 3) Successful infusion of PTCy-MILs; 4) The absence of grade III-IV acute graft-versus-host-disease (GVHD) for 90 days after PTCy-MILs infusion. Acute GVHD is defined by the Modified Keystone Criteria.

SECONDARY OUTCOMES:
Optimal safe dose for PTCy-MILs | 90 days
  Optimal safe dose is defined as the maximal MILs cell dose that can be expanded in at least 70% of patients at which upon administration does not exacerbate grade III/IV GVHD
Immunologic characterization of the PTCy-MIL product before and after expansion | up to 3 years
  Amount of MILs with expression of CD3, CD4, Cd8, CXCR4, CD45RO, CD62L, CD107a, FasL, markers of exhaustion and T-cell inactivation as identified by multi-color flow cytometry and functional studies of alloMILs and T-cell response.
Number of participants who experience chronic GVHD | up to 2 years post-transplant
  Chronic GVHD is defined by National Institutes of Health (NIH) criteria.
Clinical Response | up to 3 years
  Number of participants with complete remission (CR), partial remission (PR) and stable disease (SD) as assessed by bone marrow examination, CBC with differential, serum chemistries, cytogenetics and disease-specific molecular studies
Progression-Free Survival | up to 3 years
  Time from day of PTCy-MILs infustion to progression/relapse of disease or death from any cause, whichever occurs first
Overall Survival | up to 3 years
  Time alive from the day of PTCy-MILs infusion to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Philip Imus, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No